CLINICAL TRIAL: NCT04181476
Title: Efficacy Evaluation of Products Against Long Wavelength Ultraviolet A1 and Visible Light Induced Biological Effects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Director of Investigator-Initiated Trials, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13223
Record Dates: First submitted 2019-10-23; First posted 2019-11-29 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Sun Damaged Skin
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical products and Untreated areas (Other): The subject will serve as their own control. Four different products will be tested.
  Interventions: Drug: Sunscreening Agents

INTERVENTIONS:
Drug: Sunscreening Agents — Four different sunscreens

SUMMARY:
The purpose of this study is to evaluate the efficacy of topical products in providing protection against the visible light and ultraviolet A1 (UVA1) part of sunlight. Ultraviolet radiation and visible light are both components of sunlight that reach the earth. It is important to test these topical products against visible light and UVA1 because our current sunscreens may not protect against these very well.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 and older
* Patients Fitzpatrick skin phototype (SPT) III-IV with normal skin health
* Patient able to understand requirements of the study and risks involved

Exclusion Criteria:

* A recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post inflammatory hyperpigmentation
* A history of a relevant skin condition on any part of the patient's body (e.g. atopic dermatitis, eczema, vitiligo, sun burn, etc.
* A known history of photodermatoses
* A known history of photosensitivity disorders
* A known history of melanoma or non-melanoma skin cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in Investigator's Global Assessment (IGA) | through study completion, an average of 1 week
  Assesses erythema and pigmentation
Change in Colorimetry | through study completion, an average of 1 week
  Measures erythema and pigmentation
Change in Diffuse Reflectance Spectroscopy | through study completion, an average of 1 week
  Measures erythema and pigmentation

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, MD, Principal Investigator — Henry Ford HS
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No